CLINICAL TRIAL: NCT04681846
Title: Results of the Staged Surgical Approach for Management of Infected Un-united Femoral Shaft Fractures in Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Girgis Waheeb Tawfeek, Orthopaedic Surgeon, Assiut University
Other Study IDs: Fracture-related infection
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Fracture Non Union
Keywords: infected non-union
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Staged approach using antibiotic-cement impregnated PMMA spacer — It will be prepared in the following manner. the cement will be mixed with vancomycin in a ratio of 2 gm to each 40 gm of the spacer. The spacer should be shaped into a cylinder before its solidification. The spacer should be as big as possible to fill the whole defect, without compromising the soft tissue and skin closure. Also, cement should wrap the two ends of bone extremities on 2 or 3 centimeters.

SUMMARY:
Assessment of the efficacy of the multistage technique in the eradication of infection and achieving the union of traumatic infected femoral un-united shaft fractures in adult patients for one year follow up.

DETAILED DESCRIPTION:
All cases will be treated by the induced membrane technique in two stages. In the first stage, thorough debridement of the infected bone and soft tissues and copious lavage will be done.

After radical debridement, primary fixation will be done by either external fixation or antibiotic cement coated internally fixed implants.If there is a bone defect, it will be measured and filled with an antibiotic-impregnated (PMMA) cement spacer. The second stage procedure will be performed 4 to 8 weeks after the first one if soft tissue permits and only if there is no clinical or biochemical evidence of ongoing infection as indicated by normal white blood cell count, C-reactive protein, and erythrocyte sedimentation rate. It includes the exchange of the antibiotic cement spacer by a cancellous bone graft.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old.
2. Type 32 according to Arbeitsgemeinschaft für Osteosynthesefragen classification in adults.

Exclusion Criteria:

1. Patients with deficient soft tissue coverage with exposed bone.
2. Patients with reflex sympathetic dystrophy.
3. Spinal injuries associated with neurological complications affecting the lower limbs.
4. Associated head injury affecting the conscious level or the motor power of the injured limb.
5. Associated mutilating limb injury or peripheral amputation.
6. Bone defect more than 6 cm in length.
7. Chronic peripheral ischemia of the limb.
8. Past history of pathological fractures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient attending the department of orthopedics and traumatology, Assiut university with traumatic infected un-united femoral fractures.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in the patient-reported clinical outcome as assessed using the WOMAC Osteoarthritis Index from enrollment to 1-year follow-up after the definitive stage. | from enrollment to one year follow up after the definitive stage.
  WOMAC is composed of 24 items over 3 subscales (5 for pain, 2 for stiffness, and 17 for physical function). Participants can rate their difficulty for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Waheeb, Msc ortho, Principal Investigator — Assiut University , 71515 Assiut, Arab Republic of Egypt.; Osama Farouk, MD ortho, Study Chair — Assiut University , 71515 Assiut, Arab Republic of Egypt.; Hossam MA Abubeih, MD ortho, Study Director — Assiut University , 71515 Assiut, Arab Republic of Egypt.; Mahmoud Badran, MD ortho, Study Director — Assiut University , 71515 Assiut, Arab Republic of Egypt.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prasarn ML, Ahn J, Achor T, Matuszewski P, Lorich DG, Helfet DL. Management of infected femoral nonunions with a single-staged protocol utilizing internal fixation. Injury. 2009 Nov;40(11):1220-5. doi: 10.1016/j.injury.2009.06.009. Epub 2009 Jul 7. PMID 19586625
- [Background] Kinik H, Karaduman M. Cierny-Mader Type III chronic osteomyelitis: the results of patients treated with debridement, irrigation, vancomycin beads and systemic antibiotics. Int Orthop. 2008 Aug;32(4):551-8. doi: 10.1007/s00264-007-0342-9. Epub 2007 Mar 21. PMID 17375299
- [Background] Campoccia D, Montanaro L, Arciola CR. The significance of infection related to orthopedic devices and issues of antibiotic resistance. Biomaterials. 2006 Apr;27(11):2331-9. doi: 10.1016/j.biomaterials.2005.11.044. Epub 2005 Dec 20. PMID 16364434
- [Background] Liporace FA, Yoon RS, Frank MA, Gaines RJ, Maurer JP, Polishchuk DL, Choung EW. Use of an "antibiotic plate" for infected periprosthetic fracture in total hip arthroplasty. J Orthop Trauma. 2012 Mar;26(3):e18-23. doi: 10.1097/BOT.0b013e318216dd60. PMID 21804411
- [Background] Ohtsuka H, Yokoyama K, Higashi K, Tsutsumi A, Fukushima N, Noumi T, Itoman M. Use of antibiotic-impregnated bone cement nail to treat septic nonunion after open tibial fracture. J Trauma. 2002 Feb;52(2):364-6. doi: 10.1097/00005373-200202000-00025. No abstract available. PMID 11835003
- [Background] Micev AJ, Kalainov DM, Soneru AP. Masquelet technique for treatment of segmental bone loss in the upper extremity. J Hand Surg Am. 2015 Mar;40(3):593-8. doi: 10.1016/j.jhsa.2014.12.007. Epub 2015 Jan 31. PMID 25648786
- [Background] Masquelet AC. Induced Membrane Technique: Pearls and Pitfalls. J Orthop Trauma. 2017 Oct;31 Suppl 5:S36-S38. doi: 10.1097/BOT.0000000000000979. PMID 28938390
- [Background] Blum AL, BongioVanni JC, Morgan SJ, Flierl MA, dos Reis FB. Complications associated with distraction osteogenesis for infected nonunion of the femoral shaft in the presence of a bone defect: a retrospective series. J Bone Joint Surg Br. 2010 Apr;92(4):565-70. doi: 10.1302/0301-620X.92B4.23475. PMID 20357336
- [Background] Phillips JR, Trezies AJ, Davis TR. Long-term follow-up of femoral shaft fracture: Relevance of malunion and malalignment for the development of knee arthritis. Injury. 2011 Feb;42(2):156-61. doi: 10.1016/j.injury.2010.06.024. PMID 20656289
- [Background] Stannard JP, Bankston L, Futch LA, McGwin G, Volgas DA. Functional outcome following intramedullary nailing of the femur: a prospective randomized comparison of piriformis fossa and greater trochanteric entry portals. J Bone Joint Surg Am. 2011 Aug 3;93(15):1385-91. doi: 10.2106/JBJS.J.00760. PMID 21915543
- [Background] Weam F, El-sayed M, Mohamed M. Induced Membrane (Masquelet) Technique for Treatment of Long Bone De-fects. The Medical Journal of Cairo University 2018;86:215-222.
- [Background] Dhanasekhar R, Jacob PJ, Francis J. Antibiotic cement impregnated nailing in the management of infected non-union of femur and tibia. Kerala J Orthop 2013;26:93-97.
- [Background] Cierny G, Mader J. The surgical treatment of adult osteomyelitis. In: Evarts C. Surgery of the Musculoskeletal System, New York, USA: Churchill Livingstone; 1983; 4814-34.